CLINICAL TRIAL: NCT06781957
Title: Pharmacokinetics of Follicle-stimulating Hormone and Human Chorionic Gonadotrophin Following a Single Subcutaneous Injection of Gonadotropins-IBSA in Pituitary Down-regulated Female Subjects
Brief Title: Pharmacokinetics of FSH and hCG After a Single Subcutaneous Injection of Gonadotropins-IBSA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23CDN-FCG08
Record Dates: First submitted 2024-12-10; First posted 2025-01-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: OVARIAN STIMULATION; Infertility
Keywords: gonadotropin; FSH; hCG; infertility; Controlled ovarian stimulation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gonadotropins 75 IU (Experimental): Single dose 75 IU
  Interventions: Drug: Gonadotropins Subcutaneos
- Gonadotropins 225 IU (Experimental): Single dose 225 IU
  Interventions: Drug: Gonadotropins Subcutaneos
- Gonadotropins 450 IU (Experimental): Single dose 450 IU
  Interventions: Drug: Gonadotropins Subcutaneos

INTERVENTIONS:
Drug: Gonadotropins Subcutaneos — Gonadotropins s.c. single dose

SUMMARY:
The objectives of this study is to evaluate the PK and the dose-proportionality of FSH and HCG following a single dose of Gonadotropins-IBSA, administered subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Female of childbearing potential, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥18 and ≤45 years of age, with BMI >18.5 and <32.0 kg/m2 and body weight ≥45.0 kg.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Use of a COC containing at least 20 µg of ethinyl estradiol for at least 3 months prior to screening and willing to keep using the same oral contraceptive until the end of the study. The usual regimen (with hormone-free interval or continuous dosing) will be allowed until Day -1. Subjects must agree to take the COC in a continuous manner (no hormone-free interval) from Day 1 to Day 72.
4. Females who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized for atleast 3 months prior to dosing) must be willing to use a male condom with intravaginally applied spermicide or total abstinence from heterosexual intercourse (when this is in line with the preferred and usual lifestyle of the subject) from screening and throughout the study and for 30 days after the last study drug administration.
5. Able to understand the study procedures and provide signed informed consent to participate in the study

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening.
2. Clinically significant abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody at screening.
3. Positive pregnancy test or lactating subject.
4. Positive urine drug screen, urine cotinine test, or alcohol breath test.
5. Known allergic reactions to FSH, hCG, other gonadotropins, or other related drugs, or to any excipient in the formulation.
6. Clinically significant ECG abnormalities or vital signs abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
7. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
8. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
9. Hemoglobin <125 g/L, or hematocrit <0.32 L/L at screening.
10. FSH levels > 4 IU/L at admission in each period.
11. Clinically significant history of an abnormal menstrual cycle
12. Abnormal Pap smear prior to administration of the study drug (result is valid for 12 months).
13. History of ovarian cysts or enlargement.
14. History or presence of polycystic ovary syndrome.
15. Presence of undiagnosed vaginal and/or urinary tract bleeding.
16. History or presence of sex hormone dependent tumors of reproductive tract and accessory organs.
17. History of hypothalamus or pituitary gland tumors.
18. Personal history or strong family history (first degree relative) of coagulation disorders such as thromboembolic diseases (e.g., thrombophlebitis, pulmonary embolism or coagulation factors deficiency).
19. History of rare hereditary galactose and/or lactose intolerance (e.g., congenital lactase deficiency [CLD] or glucose-galactose malabsorption [GGM]).
20. Tattoos covering the potential study drug injection site or any skin conditions that would prevent the injection (e.g., psoriasis, major scar, etc.).
21. Use of medications for the timeframes specified below, except for the subject's prescribed COC and medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    1. depot injection or implant of any drug within 3 months prior to study drug administration.
    2. prescription medications within 14 days prior to study drug administration;
    3. any vaccine, including COVID-19 vaccine, within 14 days prior to study drug administration;
    4. over-the-counter (OTC) products and natural health products (including herbal remedies such as St. John's wort, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to study drug administration, with the exception of the occasional use of acetaminophen (up to 2 g daily);
22. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
23. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
24. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Primary PK endpoints FSH | until 240 hours post dose
  Day 72: AUC0-24
Primary PK endpoints hCG | until 240 hours post dose.
  Day 72: AUC0-24
Dose-proportionality of FSH | until 240 hours post dose
  AUC (using baseline-corrected data)
Dose-proportionality of FSH | until 240 hours post dose
  Cmax (using baseline-corrected data)
Dose-proportionality of hCG | until 240h post dose
  AUC (baseline correction)
Dose-proportionality of hCG | until 240h post dose
  Cmax (baseline correction)

SECONDARY OUTCOMES:
PD endpoints of Gonadotropins-IBSA | until 240 hours post dose
  Levels of inhibin B
PD endpoints of Gonadotropins-IBSA | until 240 hours post dose
  Levels of estradiol (E2).
Adverse events (AEs) | From the signature of the Informed Consent until the end of the study
  Percentage of subjects with any AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No